CLINICAL TRIAL: NCT02550314
Title: A Phase III Study on the Regenerative Treatment of Tympanic Membrane With NPC-18 and FBG-18-multicenter,Investigator Initiated Clinical Trial
Brief Title: A Study on the Regenerative Treatment of Tympanic Membrane With NPC-18 and FBG-18
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Responsible Party: Principal Investigator, Shin-ichi Kanemaru, director, Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRIENT1328
Record Dates: First submitted 2015-09-11; First posted 2015-09-15 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Tympanic Membrane Perforation
MeSH Terms: conditions — Tympanic Membrane Perforation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NPC-18,FBG-18 (Experimental): Intervention drug:
  NPC-18;trafermin(recombination) and gelatin spnge, combination drug FBG-18;fibrin glue
  Usage:NPC-18 and FBG-18 is administered at the same time for regenerative treatment of tympanic membrane
  Interventions: Drug: fiblast,gelatin sponge,fibrin glue

INTERVENTIONS:
Drug: fiblast,gelatin sponge,fibrin glue

SUMMARY:
To assess the efficacy and safety of the regeneration treatment of tympanic membrane with NPC-18 and FBG-18.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed concent obtained
2. At the time of obtaining informed consent, Ages ranged from over 20 to 80
3. At the time of obtaining informed consent, only those with tympanic membrane perforation in 1 ear (not both) for over 6 months (perforation in both ears is excluded)

Exclusion Criteria:

1. TMP caused by burn or radiation therapy
2. In patients with chronic otitis media with ear drum perforation, tympanic cavity are not dry
3. Inflammatory,infection or otorrhea in patient's eardrum,earcanal,middle ear and tympanic cavity
4. No invasion of epithelial and no cholesteatoma in tympanic cavity or around perforated edge
5. History of tympanoplasty
6. A Part of the eardrum adhered to tympanic cavity
7. By temporal bone CT, soft tissue shadow in mastoid antrum or tympanic (using a CT image of less than 12 wks before patients registration)
8. Abnormality in the chain and ear ossicles
9. Air-bone gap difference more than 25dB by patch hearing test
10. Unable to see whole edge of TMP due to narrow external auditory canal
11. Unable to wash out Ear drops during the treatment period
12. Presenting with uncontrolled diabetes (NGSP HbA1c 6.9% and more)
13. Presenting with autoimmune disease
14. History of malignancy within 3 years prior to obtained informed concent
15. Administration of immunosuppressive agent or anti-cancer-agent
16. History of Allergic reaction to local anesthetic(Xylocaine), bFGF(Fiblast spray), fibrin glue(Beriplast P Combi set, etc.), gelatin sponge formulation(spongel) and others
17. Though out the period from screening to treatment, patient who is unable to wash out "Thrombolytic agent", "Anticoagulant", "Anti-platelet agent", "Procoagulant agent", "anti-line solvent"and"aprotinin formulation"

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Closure of tympanic membrane perforation in the observation period at16 wks | Closure of tympanic membrane perforation in the observation period at16 wks

SECONDARY OUTCOMES:
Closure of tympanic membrane perforation in the observation period at 4 wks | Closure of tympanic membrane perforation in the observation period at 4 wks
Improvement of hearing level in the observation period at 4 wks and 16 wks | Improvement of hearing level in the observation period at 4 wks and 16 wks
Air-bone gap in the observation period at 4 wks and 16 wks | Air-bone gap in the observation period at 4 wks and 16 wks
The difference of the average hearing level of air conduction threshold from the treatment at 0 wk and observation period at 4wks and 6 wks | The difference of the average hearing level of air conduction threshold from the treatment at 0 wk and observation period at 4wks and 6 wks
Average hearing level of air conduction threshold in the observation period at 4 wks and 16 wks | Average hearing level of air conduction threshold in the observation period at 4 wks and 16 wks

IPD SHARING:
Plan to Share IPD: Undecided